CLINICAL TRIAL: NCT02406066
Title: Phase 1 Combined Single and Multiple Rising Dose Study of the Safety and Pharmacokinetics of Metyrapone/Oxazepam Combination (EMB-001)
Brief Title: Single and Multiple Rising Dose Study of Safety and PK of Metyrapone/Oxazepam Combination (EMB-001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Embera NeuroTherapeutics, Inc. (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ERL-001; 5R01DA030932-04 (NIH)
Record Dates: First submitted 2014-04-16; First posted 2015-04-02 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2016-07

CONDITIONS: Cocaine Use Disorder; Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Metyrapone; Oxazepam; KPNA1 protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Subjects will receive capsules containing no active pharmaceutical ingredients.
  Interventions: Drug: Placebo
- Low Dose (Cohort 1) (Active Comparator): 270 mg metyrapone and 12 mg oxazepam, given once for the single-dose phase of the study, followed by BID dosing for approximately one week
  Interventions: Drug: metyrapone & oxazepam
- Medium Dose (Cohort 2) (Active Comparator): 540 mg metyrapone and 24 mg oxazepam, given once for the single-dose phase of the study, followed by BID dosing for approximately one week
  Interventions: Drug: metyrapone & oxazepam
- High Dose (Cohort 3) (Active Comparator): 720 mg metyrapone and 24 mg oxazepam, given once for the single-dose phase of the study, followed by BID dosing for approximately one week
  Interventions: Drug: metyrapone & oxazepam

INTERVENTIONS:
Drug: metyrapone & oxazepam — 6 subjects will receive active study drug (a low dose combination of metyrapone & oxazepam) and 2 subjects will receive placebo.
  Other Names: Cohort 1
  Arms: Low Dose (Cohort 1)
Drug: metyrapone & oxazepam — 6 subjects will receive active study drug (a medium dose combination of metyrapone & oxazepam) and 2 subjects will receive placebo.
  Other Names: Cohort 2
  Arms: Medium Dose (Cohort 2)
Drug: metyrapone & oxazepam — 6 subjects will receive active study drug (a high dose combination of metyrapone & oxazepam) and 2 subjects will receive placebo.
  Other Names: Cohort 3
  Arms: High Dose (Cohort 3)
Drug: Placebo — Each cohort will have 2 subjects receiving placebo
  Other Names: All Cohorts
  Arms: Placebo

SUMMARY:
This is a study of EMB-001 (a combination of two FDA-approved drugs, metyrapone and oxazepam) in otherwise healthy adults who are regular cigarette smokers. There will be 3 groups of 8 subjects; in each group, 6 subjects will get the drug combination and 2 will get placebo. Neither the subjects nor the study personnel will know who got drug and who got placebo (double-blind). In the first group the drug doses will be low, and they will be increased in the second and third groups. Subjects will receive a single dose on Day 1, followed 24 hours later by the start of doses twice daily for 7 days, and then a final morning dose on the last day. The levels of the drugs in the blood will be assessed by repeated blood draws after the first day and after the end of dosing. Safety will be assessed after the single dose and repeated dosing. Effects of study drug on smoking and craving cigarettes will be assessed at the end of repeated dosing. The hypothesis is that this drug combination will be safe, with relatively few side effects.

DETAILED DESCRIPTION:
This study is a Phase 1, double blind, single and multiple rising dose tolerance study of EMB-001 (metyrapone/oxazepam combination) in otherwise healthy adults who have tobacco use disorder. There will be 3 cohorts, each with 8 subjects (6 active: 2 placebo), for a total of 24 subjects. During the treatment period, subjects will receive a single dose of EMB 001 on Day 1, followed 24 hours later by the start of multiple doses twice daily for 7 days, and then a final morning dose on the last dosing day (Day 9). This design allows for characterization of EMB-001 single dose PK for 24 hours, followed by assessment of repeat dose PK in the multiple-dose phase. Safety will be assessed after the single dose and repeated dosing. Effects of study drug on smoking and craving cigarettes will be assessed at the end of repeated dosing. Later studies may also assess the efficacy of this drug combination in treating cocaine use disorder, tobacco use disorder, and/or other disorders.

ELIGIBILITY:
Inclusion Criteria:

* Males and females of Non-Childbearing Potential age 18-65
* Have provided written informed consent prior to any study procedures
* Are willing and able to comply with all aspects of the protocol
* Normal or clinically acceptable screening electrocardiogram (ECG)
* Normal blood pressure (systolic: 90-140 mmHg; diastolic 50-90 mmHg) and heart rate (50-100 bpm)
* Smoke at least 10 cigarettes per day (for approximately 1 year or longer)
* Body mass index > 18.5 and < 35

Exclusion Criteria:

* Known hypersensitivity to or intolerance of oxazepam or metyrapone, or any benzodiazepine
* Subjects with a low out-of-range serum cortisol value at screening or subjects who, in the investigator's opinion, have a heightened likelihood of having adrenal insufficiency.
* Subjects who have a positive urine drug screen for illegal drugs or other drugs with a high potential for abuse (other than nicotine).
* Inability to communicate or cooperate with the investigator
* History of drug dependence (except nicotine) or psychiatric illness within the past 2 years.
* Subjects with any history of adrenal insufficiency or other adrenal, hypothalamic, or pituitary disorders.
* History of asthma or other respiratory disease, neurologic or neuromuscular disease, or hypotension or cardiovascular disease, that may, in the opinion of the investigator, impact any study procedures or measures, or compromise the safety of the subject.
* Other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results and, in the judgment of the Investigator or Sponsor, would make the subject inappropriate for entry into this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-03; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Safety/Tolerability based on multiple safety parameters (adverse events (AE), physical examinations, vital signs, 12-lead ECG, Sheehan Suicidality Tracking Scale (S STS) and laboratory tests) | Daily on Days 1-12, and on Day 17. Study Completion occurs on Day 17.
  Safety will be assessed through monitoring of adverse events (AE), physical examinations, vital signs, 12-lead ECG, Sheehan Suicidality Tracking Scale (S STS) and laboratory tests.

SECONDARY OUTCOMES:
Pharmacokinetics (Plasma PK parameters will be serially assessed for oxazepam, metyrapone, and for the primary metabolite of metyrapone, metyrapol) | After single- and multiple-dosing- Samples will be drawn on Day 1 and Day 10 at the following times Pre-dose, .25, .5, .75, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 36, & 48 hours.
  Plasma PK parameters will be serially assessed for oxazepam, metyrapone, and for the primary metabolite of metyrapone, metyrapol.

OTHER OUTCOMES:
Craving/addiction measures | These will be assessed at baseline and on Study Day 9
  Exploratory efficacy endpoints will include the following craving and addiction measures:
  1. The Smoking Urges Questionnaire-Brief
  2. Minnesota Nicotine Withdrawal Scale
  3. Number of cigarettes smoked, breath carbon monoxide, and urine cotinine.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Connor, RN, Study Director — Embera NeuroTherapeutics, Inc.
Locations (2):
- United States (2):
  - Collaborative Neuroscience Network, LLC, Long Beach, California
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana

REFERENCES:
- See also: Sponsor: Embera NeuroTherapeutics — http://www.emberaneuro.com/